CLINICAL TRIAL: NCT02520024
Title: Assessing the Impact of Self-directed Care, Within a Medicaid-funded Environment,on Participation and Community Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University Collaborative on Community Inclusion (Other)
Responsible Party: Principal Investigator, Mark Salzer, Director, Temple University Collaborative on Community Inclusion
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 13304
Record Dates: First submitted 2015-08-01; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Major Depression; Bipolar Disorder; Schizophrenia
Keywords: self-directed care; serious mental illness
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-directed Care (Experimental): Individuals in the experimental condition will work with a specially trained certified peer specialists (CPS) who will serve as "recovery coaches" to develop an individualized recovery plan that describes their goals and desires. They will then work with the team to select both the behavioral health treatment and rehabilitation services, and the non-behavioral health materials and resources they believe are necessary to achieve their goals.
  Interventions: Behavioral: self-directed care
- Treatment as usual (No Intervention): Participants in the control condition will receive services as usual.

INTERVENTIONS:
Behavioral: self-directed care
  Arms: Self-directed Care

SUMMARY:
This project proposed to demonstrate the effectiveness, costs, and benefits to participation and community living self-directed care programming within a financially sustainable Medicaid managed care environment. The study examined outcomes associated with the implementation of a novel self-directed care (SDC) approach being implemented in Delaware County, Pennsylvania in which consumers were able to access a set amount of renewable funds per year and direct how they were spent, both to purchase the types and amounts of rehabilitation and treatment services they desire (and from whom they choose) and to purchase a broad-range of individualized resources and services that are generally outside of Medicaid funding (e.g., health club memberships, yoga classes, support in taking care of bills).

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18-65 who are currently receiving Medicaid-reimbursed services in Delaware County, Pennsylvania for either a schizophrenia-spectrum, major depression, or bipolar disorder;
2. Individuals with a cost profile within the 60-90% band of all Magellan-administered Medicaid recipients in the county (estimated service costs between $10,048 and $22,324); 3) No more than two inpatient hospitalizations of 10 days per stay, over a 2 year period prior to the study;

4) No hospitalization within 6 months of the study; 5) Ability to understand self-directed care requirement and express interest in working with a "recovery coach."

Exclusion Criteria:

1. do not speak English;
2. have a legal guardian;
3. are unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline TU Community Participation Questionnaire to follow up at 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
  Used to gather information about the frequency of participation in multiple domains (e.g., employment, education, spirituality, leisure/recreation, attendance at self-help groups, etc.) in the last 30 days, whether or not they did the activity enough, not enough, or too much in addition to their level of satisfaction with their level of participation in the activity.
Change from Baseline Recovery Assessment Scale to follow up at 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
Change from Baseline Quality of Life to 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
Change from Baseline Hopkins Symptom Checklist to 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
Change from Baseline Empowerment Scale to 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
Change from Baseline Coping Mastery Questionnaire to 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
Change from Baseline Perceived Competence for Recovery Questionnaire to 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
Change from Baseline Perceived Autonomy Support: The Mental Health Questionnaire to 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
Change from Baseline Elements of a Recovery Facilitating Systems Assessment Questionnaire - Adult Version to 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
Change from Baseline Revised Camberwell Assessment of Need Questionnaire to 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline
Change from Baseline Treatment Self-Regulation Questionnaire to 12 months and 24 months post-baseline | Baseline, 12 months- and 24 months post-baseline